CLINICAL TRIAL: NCT03152708
Title: The Exploratory Study on CAN008 Biomarker CD95 Ligand and Its Promoter (CpG2) Methylation in Chinese Patients With Glioblastoma
Brief Title: CAN008 Biomarker CD95 Ligand and CpG2 Methylation in Chinese Patients With Glioblastoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: CANbridge Life Sciences Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CAN-B1-008-L-009
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was conducted on the post-operative tumor tissues from 62 GBM patients. 20 slices are necessary for all the CD95 and CpG2 test in the central lab by the methods of immunisation and DNA methylation.

ELIGIBILITY:
Inclusion Criteria:

* Chinese nationality
* No limits on Gender and age
* First diagnosed GBM
* Brain tumor tissue cytological diagnosis of glioblastoma (GBM, pleomorphic glioblastoma, WHO level IV)

Exclusion Criteria:

* Other types of glioma by histological diagnosis
* Tumor tissue not eligible for the central laboratory testing standard
* No enough tumor tissue for the central laboratory test

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese GBM patients
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2017-11-01 (Estimated); Primary Completion 2017-12-01 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
CD95 Ligand Positive Rate | 0 day

SECONDARY OUTCOMES:
CpG2 Positive Rate | 0 day

CONTACTS AND LOCATIONS:
Overall Officials: Jinsong Wu, MD, Principal Investigator — Huashan Hospital

IPD SHARING:
Plan to Share IPD: No